CLINICAL TRIAL: NCT02534454
Title: Transcranial Direct Current Stimulation (TDCS) and Cognitive Retraining to Augment Pharmacotherapy for the Treatment of Nicotine Dependence
Brief Title: TDCS and Cognitive Retraining to Augment Pharmacotherapy for the Treatment of Nicotine Dependence
Acronym: TDCSNIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Mind Research Network (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 20547; R21DA037546 (NIH)
Record Dates: First submitted 2015-08-24; First posted 2015-08-27 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine Replacement Therapy; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active TDCS + Active Retraining (Experimental): 2.0 milliamperes (mA) of transcranial direct current stimulation (TDCS) applied during active nicotine avoidance retraining
  Interventions: Behavioral: Active Retraining; Device: Active transcranial direct current stimulation (TDCS); Drug: Nicotine Replacement Therapy (Habitrol)
- Sham TDCS + Active Retraining (Experimental): 0.1 mA of transcranial direct current stimulation (TDCS) applied during active nicotine avoidance retraining
  Interventions: Behavioral: Active Retraining; Device: Sham transcranial direct current stimulation (TDCS); Drug: Nicotine Replacement Therapy (Habitrol)
- Active TDCS + Sham retraining (Experimental): 2.0 mA of transcranial direct current stimulation (TDCS) applied during sham nicotine avoidance retraining
  Interventions: Behavioral: Sham Retraining; Device: Active transcranial direct current stimulation (TDCS); Drug: Nicotine Replacement Therapy (Habitrol)
- Sham TDCS + Sham Retraining (Experimental): 0.1 mA of transcranial direct current stimulation (TDCS) applied during sham nicotine avoidance retraining
  Interventions: Behavioral: Sham Retraining; Device: Sham transcranial direct current stimulation (TDCS); Drug: Nicotine Replacement Therapy (Habitrol)

INTERVENTIONS:
Behavioral: Active Retraining
  Arms: Active TDCS + Active Retraining; Sham TDCS + Active Retraining
Behavioral: Sham Retraining
  Arms: Active TDCS + Sham retraining; Sham TDCS + Sham Retraining
Device: Active transcranial direct current stimulation (TDCS)
  Arms: Active TDCS + Active Retraining; Active TDCS + Sham retraining
Device: Sham transcranial direct current stimulation (TDCS)
  Arms: Sham TDCS + Active Retraining; Sham TDCS + Sham Retraining
Drug: Nicotine Replacement Therapy (Habitrol) — Administration of Nicotine Replacement Therapy Patches

SUMMARY:
The purpose of the phase 1 translational pilot study proposed here is to gather preliminary data investigating the efficacy of transcranial direct current stimulation (TDCS) and cognitive retraining to enhance nicotine replacement therapy for smoking cessation. The recent use of TDCS over task relevant regions to alter behavior holds incredible promise for use in cognitive retraining intervention protocols. Previous studies of cognitive retraining have focused on implicit training techniques. This proposed study will attempt to enhance these implicit training techniques through the use of TDCS during implicit retraining in order to increase learning of avoidance-related action tendencies towards tobacco. The objective of this pilot study is to establish the feasibility and obtain preliminary data on the effectiveness of using brain stimulation with cognitive retraining to reduce cigarette smoking in individuals with nicotine addiction.

ELIGIBILITY:
Inclusion Criteria:

* Consume 10 or more cigarettes/day average for the past 60 days
* Able to provide informed consent
* Less than 3 months smoking abstinence in the past year
* Right Handed

Exclusion Criteria:

* Serious medical illness within 6 months (e.g. cancer, hepatic, or renal disease)
* Significant cardiovascular disease (e.g. recent stroke or heart attack, arrhythmias, worsening angina pectoris, uncontrolled hypertension) generalized skin disorders, or sensitivity to the nicotine patch
* Use of illicit drugs (excluding marijuana) in the previous 30 days
* Psychosis, psychotic disorder, or bipolar disorder
* Current active major depression (depressive episode within last month)
* Clinically significant suicidal ideation
* Prior seizure
* Current bupropion or tricyclic antidepressants
* Current pregnancy, trying to become pregnant, or breastfeeding
* Current active alcohol dependence (symptoms in last 30 days)
* Left-handedness
* Current medication known to interact with nicotine replacement therapy (NRT) or smoking cessation (e.g. adenosine, cimetidine, conivaptan, cyproterone, peginterferon alfa-2bg, tocilizumab, theophylline)
* Metal in the head
* Implanted brain medical devices
* Electromedical devices
* Latex Allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2015-08-15 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Cigarettes per Smoking Day | 11-Weeks Post-transcranial direct current stimulation (TDCS)/Retraining
  Number of cigarettes consumed per day will be assessed using the Timeline Follow-back method to obtain the number of cigarettes consumed on each day since the last administration of the Timeline Follow-back. Cigarettes per smoking day will be the mean number of cigarettes consumed on days on which cigarettes were consumed.

SECONDARY OUTCOMES:
Approach Bias Towards Cigarettes (Measure of response time differences) | 1 week Post-transcranial direct current stimulation (TDCS)/Retraining
  Measure of response time differences to push vs. pull a joystick in response to pictures of cigarettes vs. control objects (e.g. pens)

CONTACTS AND LOCATIONS:
Locations (1):
- The Mind Research Network, Albuquerque, New Mexico, United States